CLINICAL TRIAL: NCT06246123
Title: Post Marketing Surveillance of Jyseleca Tab. (Filgotinib Maleate) in Korean Subjects
Brief Title: A Study of Jyseleca Tablet (Filgotinib Maleate) in Korean Participants
Status: Recruiting | Type: Observational
Sponsor: Eisai Korea Inc. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: FIL-M082-501
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Arthritis, Rheumatoid; Colitis, Ulcerative
Keywords: Filgotinib Maleate; Rheumatoid arthritis; Ulcerative colitis; FIL-M082-501
MeSH Terms: conditions — Arthritis, Rheumatoid; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: Korean participants who are prescribed with Jyseleca (Filgotinib Maleate) tablet 100 mg and 200 mg per approved prescribing information of Filgotinib Maleate in the post marketing setting will be enrolled and observed for up to 24 weeks or until discontinuation of treatment due to AEs or any other reason, whichever occurs first.
  Interventions: Other: Non-interventional

INTERVENTIONS:
Other: Non-interventional — No intervention will be administered.

SUMMARY:
The purpose of this study is to collect and evaluate the following information in relation to the safety and the efficacy of Jyseleca tablet (Filgotinib Maleate) 100 milligram (mg) and 200 mg in this post marketing setting: (1) Serious adverse events and adverse drug reactions (2) Unexpected adverse events and adverse drug reactions not reflected in precautions for use (3) Known adverse drug reactions (4) Non-serious adverse events and adverse drug reactions (5) Other safety and effectiveness related information will be evaluated in accordance with the permitted articles under the actual conditions of use in Korea.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who are being administered with Jyseleca tablet in accordance with the Korean approved label therapeutic indications.

* Korean local label therapeutic indications of Jyseleca tablet. In the following participants, Jyseleca tablet should be used only if they do not respond appropriately or are intolerant to existing treatments.
* Following:

  1. Participants over 65 years of age.
  2. Participants with a high cardiovascular risk.
  3. Participants with malignancy.
* Rheumatoid arthritis:

  1. For treatment of moderately to severely active rheumatoid arthritis in adults who have responded inadequately to, or who are intolerant to one or more disease-modifying anti-rheumatic drugs (DMARDs).
  2. Jyseleca tablet may be used as monotherapy or in combination with methotrexate (MTX).
  3. Jyseleca tablet should not be used in combination with biological DMARDs (bDMARDs) or other Janus kinase (JAK) inhibitors.
* Ulcerative colitis:

  a. For treatment of moderately to severely active ulcerative colitis in adults who have an inadequate response with, lost response to, or were intolerant to either conventional therapy (corticosteroids, immunosuppressants, etc.) or biological agents.
* The investigator should refer to local label and contraindications in Korea regarding the inclusion criteria.

Exclusion Criteria:

1. Individuals who fall under contraindications to the administration of Jyseleca tablet in accordance with the local label by the medical judgment of the investigator.

   * Contraindication for Jyseleca tablet in accordance with the Korean label:

     1. Participants with hypersensitivity to the active ingredient or other ingredients of the Jyseleca tablet.
     2. Participants with active infections, including serious (example, sepsis) or local infections.
     3. Participants with active tuberculosis.
     4. Participants with severe hepatic disorder.
     5. Participants with end-stage renal disorder.
     6. Participants with absolute neutrophil count (ANC) <1*10^9 cells/liters (L)
     7. Participants with absolute lymphocyte count (ALC) <0.5*10^9 cells/L
     8. Participants with hemoglobin level <8 grams per deciliter (g/dL)
     9. Pregnant or potentially pregnant women, lactating women
     10. Jyseleca tablet should not be administered to participants with genetic problems such as galactose intolerance, total lactase deficiency, or glucose-galactose malabsorption as it contains lactose.
2. Individuals who are administered Filgotinib in a clinical study other than this post marketing surveillance.
3. Individuals who are considered incompatible with participate in this surveillance by the medical judgment of the investigator.

   * The investigator should refer to local label and contraindications in Korea regarding the exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korean participants who are prescribed with Jyseleca (Filgotinib Maleate) tablet 100 mg and 200 mg per the approved prescribing information will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 2040 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Serious Adverse Events (SAEs) | From the date of enrollment up to 24 weeks
  A SAE is defined as any undesirable medical occurrence: resulting in death; life threatening; requiring hospitalization or extension of hospitalization; resulting in persistent or significant disability or functional impairment; resulting in congenital malformation or abnormality or other medically significant events than above mentioned criteria.
Number of Participants With Adverse Drug Reactions (ADRs) | From the date of enrollment up to 24 weeks
  An ADR is defined as harmful and unintended reaction to the proper administration/use of drugs, in which a causal relationship with the drug in question cannot be ruled out. Adverse events (AEs) with unknown causality to the drug among those voluntarily reported will be also considered ADRs.
Number of Participants With Unexpected AEs | From the date of enrollment up to 24 weeks
  An unexpected AE is an AE with a difference in nature, severity, specificity, or outcome, which have not been mentioned in the product licensure/safety notification of the drug.
Number of Participants With Unexpected ADRs | From the date of enrollment up to 24 weeks
  Unexpected ADR is also an unexpected AE, where unexpected AE is an AE with a difference in nature, severity, specificity, or outcome, which have not been mentioned in the product licensure/safety notification of the drug.
Number of Participants With Known ADRs | From the date of enrollment up to 24 weeks
  Known AEs are those listed in product licensure/notification of the drug and are also considered as known ADRs.
Number of Participants With Non-serious AEs | From the date of enrollment up to 24 weeks
  Non-serious AEs are other than SAE among AEs. An AE is defined as any undesirable and unintended signs (example, abnormalities in laboratory test) or symptoms/diseases occurring during administration/use of drugs, which do not need causal relationship with relevant study drug.
Number of Participants With Non-serious ADRs | From the date of enrollment up to 24 weeks
  Non-serious ADRs are other than SAE among ADR. An ADR is defined as harmful and unintended reaction to the proper administration/use of drugs, in which a causal relationship with the drug in question cannot be ruled out.
Change From Baseline in Disease Activity Score 28 Based on C-Reactive Protein (DAS28-CRP) at Week 12 and Week 24 | Baseline, Week 12 and Week 24
  The DAS28 index for rheumatoid arthritis participants was a composite score of weighted components including tender joint counts of 28, swollen joint counts of 28, participant global assessment of disease activity score, and CRP value. A DAS28-CRP score of 5.1 or above =high disease activity, a value between greater than (>) 3.2 and 5.1 =moderate disease activity and value between 2.6 and 3.2 =low disease activity, value less than (<) 2.6 =disease remission.
Change From Baseline in the Mayo Clinic Score (MCS) at Week 12 and Week 24 | Baseline, Week 12 and Week 24
  The Mayo Clinic Score for ulcerative colitis participants is comprised of 4 parts: stool frequency, rectal bleeding, endoscopic findings, and physician's global assessment, each scored from 0 to 3, where 0=normal, 3=severe. The total score ranges from 0 to 12, with higher scores indicating increased severity of disease.

CONTACTS AND LOCATIONS:
Locations (42):
- South Korea (42):
  - Site #28, Ansan
  - Site #10, Busan
  - Site #11, Busan
  - Site #15, Busan
  - Site #16, Busan
  - Site #17, Busan
  - Site #5, Busan
  - Site #7, Busan
  - Site #22, Changwon
  - Site #14, Cheongju-si
  - Site #2, Choonchen
  - Site #12, Daegu
  - Site #20, Daegu
  - Site #21, Daegu
  - Site #26, Daegu
  - Site #36, Daegu
  - Site #3, Daegu
  - Site #6, Daejeon
  - Site #9, Gwangju
  - Site #35, Gyeonggi-do
  - Site #13, Jeju City
  - Site #29, Jeonbuk
  - Site #18, Jeonju
  - Site #37, Jeonnam
  - Site #23, Jinju
  - Site #31, Kyungpook
  - Site #33, Kyungpook
  - Site #19, Seoul
  - Site #1, Seoul
  - Site #27, Seoul
  - Site #30, Seoul
  - Site #32, Seoul
  - Site #34, Seoul
  - Site #38, Seoul
  - Site #39, Seoul
  - Site #40, Seoul
  - Site #41, Seoul
  - Site #42, Seoul
  - Site #8, Seoul
  - Site #24, Wŏnju
  - Site #4, Wŏnju
  - Site #25, Yŏngin

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.
Time Frame: NOTE: IPD Sharing Time Frame has not been entered.
Access Criteria: NOTE: IPD Sharing Access Criteria has not been entered.